CLINICAL TRIAL: NCT03532191
Title: Improving the HIV PrEP Cascade Using an Intervention for Healthcare Providers
Acronym: PrEP-OI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: San Francisco Department of Public Health (Other Government); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: R01NR017573 (NIH); R01NR017573 (NIH)
Record Dates: First submitted 2018-04-29; First posted 2018-05-22 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: HIV/AIDS
Keywords: Quality Improvement; Healthcare Providers; Health Disparity
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: The proposed intervention study will be implemented using a stepped-wedge design, which is a type of one-way crossover design in which all clinics will begin the study without the PrEP-OI intervention. Each clinic will cross over to receive the intervention one-by-one every month, with the order of clinic crossover determined at random to maximize internal validity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PrEP-OI Intervention (Experimental): All clinics that have crossed over to initiate the intervention at this time. The order of crossover is determined at random.
  Interventions: Other: PrEP Optimization Intervention (PrEP-OI)
- Control until randomized for intervention (No Intervention): All clinics that have not yet initiated the intervention at this time (i.e., control clinics). A new clinic will cross over to receive the intervention each month, with the order of clinic crossover determined at random, until all clinics are receiving the intervention.

INTERVENTIONS:
Other: PrEP Optimization Intervention (PrEP-OI) — PrEP-Rx + PrEP Coordinator
  Arms: PrEP-OI Intervention

SUMMARY:
The PrEP Optimization Intervention (PrEP-OI) aims to educate healthcare providers on PrEP and assist providers in the appropriate targeting of patients at increased risk for HIV acquisition, initiating PrEP when appropriate, and providing guidance on the ongoing monitoring and adherence counseling of patients on PrEP. The intervention includes a web-based panel management tool (called PrEP-Rx) and PrEP coordination (by a PrEP Coordinator). The PrEP-OI study will take place among participating primary care and specialty clinics across the San Francisco Department of Public Health.

DETAILED DESCRIPTION:
Despite data indicating nearly 80,000 individuals starting HIV pre-exposure prophylaxis (PrEP) by the end of 2015, the Centers for Disease Control and Prevention (CDC) estimates that there are over 1.2 million adults with a substantial risk for HIV acquisition. Therefore, only 6% of these individuals are receiving PrEP. One of the barriers to PrEP implementation is lack of healthcare provider (HCP) knowledge and willingness to prescribe it. In a 2015 national survey, only 66% of primary care clinicians were aware of PrEP. However, once PrEP was defined, 91% indicated a willingness to prescribe it for high risk patients and expressed an interest in education about how to deliver PrEP. A descriptive report on the early experiences with PrEP uptake and delivery in San Francisco identified the following priority steps for HCPs to address PrEP delivery issues and to maximize PrEP's public health impact: (1) increase PrEP knowledge among HCPs and (2) expand PrEP access by training HCPs and developing tools to facilitate PrEP delivery in clinical settings. Additionally, based on the framework of the PrEP care continuum, interventions to enhance PrEP uptake include HCP education, tools to assess sexual risk, and systems to minimize HCP burden. Given these proposals and recommendations, innovative and effective approaches are needed to support and provide guidance to HCPs regardless of level of experience prescribing PrEP.

The investigators propose a PrEP optimization intervention targeted at HCPs to increase PrEP uptake and persistence among those at risk for HIV acquisition. This intervention includes: (1) an integrated web-based panel management tool called PrEP-Rx, which provides structured HIV risk assessment, automates reminders for laboratory testing and appointments, and reports patients' history of PrEP use; and (2) a centralized PrEP coordination overseen by a clinical support staff (referred to as the PrEP coordinator) who can identify individuals at high risk for HIV through direct patient contact or by reviewing registries for sexually transmitted infections (STIs) and who can support multiple HCPs. PrEP-Rx consists of three components: (a) Risk Assessment, (b) Provider Dashboard, and (c) Knowledge Base. The brief online behavioral Risk Assessment will be provided to patients to complete prior to their initial visits with HCPs. This assessment allows patients to respond to sensitive risk questions in private, removes the need for HCPs to ask detailed risk questions, provides a standardized and comprehensive view of patient's HIV risk, and decreases the time burden on HCPs. Based on responses to the Risk Assessment, a patient's risk is categorized (high, medium, or low) and results are presented to the HCP on a "Provider Dashboard" along with laboratory test results that are required prior to PrEP initiation, and the patient's history of PrEP use (if applicable). Based on these data, the HCP and patient can discuss the risks and benefits of PrEP initiation. If a PrEP prescription is given, PrEP-Rx will generate automated follow-up reminders which are sent to the PrEP Coordinator for scheduling office appointments or laboratory visits. The activities of PrEP-Rx and the role of the HCP are augmented and managed by the PrEP Coordinator, who has the ability to identify and contact patients who have tested positive for STIs, follow-up with patients to minimize loss-to-follow-up and improve adherence, and ensure timely laboratory monitoring. PrEP-Rx also contains a Knowledge Base for HCP education and ongoing training.

Therefore, the investigators propose the following aims:

Primary Aim: Evaluate the efficacy of the PrEP optimization intervention (PrEP Coordinator + PrEP-Rx) to increase PrEP prescriptions through a stepped-wedge design among 10 San Francisco primary care clinics. The investigators hypothesize that the mean number of prescriptions issued will be significantly higher when the clinics use the PrEP intervention versus when they do not.

Secondary Aims:

1. Explore differences in PrEP initiation, duration of use, and reasons for discontinuation based on patient's age, race/ethnicity, and sex/gender, and by clinic and HCP characteristics among study clinics.
2. Explore sustainability of the intervention during an eight-month follow-up after the Stepped-wedge Phase.
3. Investigate facilitators and barriers of PrEP delivery and experiences with the proposed PrEP intervention through qualitative interviews with HCPs, PrEP Coordinators, and clinic directors of study clinics.

The combination of the PrEP Coordinator plus PrEP-Rx has the potential to improve all steps of the PrEP continuum and enhance overall care by identifying individuals at high risk of HIV acquisition, standardizing HIV risk assessment, helping in PrEP initiation, systematizing follow-up visits or laboratory assessments, and educating HCPs about emerging PrEP data. These goals can have a significant public health impact and be attained with minimal burden on existing clinic resources.

ELIGIBILITY:
Inclusion Criteria:

* San Francisco Department of Public Health (DPH) clinics that have agreed to participate
* HCPs and medical directors employed at the study clinics
* Patients who are seen at these study clinics and are offered HIV PrEP during the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Efficacy of PrEP-OI | 10 months
  Mean number of PrEP prescriptions initiated

SECONDARY OUTCOMES:
PrEP usage | 10 months
  Explore differences in PrEP initiation, duration of use, and reasons for discontinuation
Sustainability during 12 month Follow-up Phase | 22 months
  Explore sustainability of the intervention by determining if prescription numbers change in the Follow-up relative to the Stepped-wedge Phase
Facilitators and barriers of PrEP delivery | 22 months
  Investigate facilitators and barriers of PrEP delivery and experiences with the proposed PrEP intervention through one-on-one qualitative interviews with HCPs and PrEP Coordinators

CONTACTS AND LOCATIONS:
Overall Officials: Parya Saberi, PharmD, MAS, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Center for AIDS Prevention Studies, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Saberi P, Stoner MCD, Ming K, Lisha NE, Hojilla JC, Scott HM, Liu AY, Steward WT, Johnson MO, Neilands TB. The effect of an HIV preexposure prophylaxis panel management strategy to increase preexposure prophylaxis prescriptions. AIDS. 2022 Nov 1;36(13):1783-1789. doi: 10.1097/QAD.0000000000003283. Epub 2022 Jun 22. PMID 35730363
- [Result] Shrestha I, Ming K, Jimenez V, Wendelborn J, Vazquez A, Steward W, Scott H, Saberi P. Lessons Learned from an HIV Pre-Exposure Prophylaxis Coordination Program in San Francisco Primary Care Clinics. AIDS Res Hum Retroviruses. 2022 Aug;38(8):611-614. doi: 10.1089/AID.2022.0013. Epub 2022 Jun 16. PMID 35592996
- [Result] Saberi P, Ming K, Shrestha I, Scott H, Thorson B, Liu A. Feasibility and Acceptability of Home-Collected Samples for Human Immunodeficiency Virus Preexposure Prophylaxis and Severe Acute Respiratory Syndrome Coronavirus 2 Laboratory Tests in San Francisco Primary Care Clinics. Open Forum Infect Dis. 2022 Jan 21;9(2):ofab657. doi: 10.1093/ofid/ofab657. eCollection 2022 Feb. PMID 35087913
- [Result] Chan CT, Ming K, Camp C, Saberi P. Sexual Behaviors, Substance Use, and Quality of Life Among Individuals Using PrEP in San Francisco During the COVID-19 Pandemic Shelter-In-Place Orders: A Cross-Sectional Survey. J Acquir Immune Defic Syndr. 2022 Apr 1;89(4):e39-e42. doi: 10.1097/QAI.0000000000002900. No abstract available. PMID 34974469
- [Result] Saberi P, Ming K, Scott H, Liu A, Steward W. "You can't have a PrEP program without a PrEP Coordinator": Implementation of a PrEP panel management intervention. PLoS One. 2020 Oct 16;15(10):e0240745. doi: 10.1371/journal.pone.0240745. eCollection 2020. PMID 33064763
- [Result] Ming K, Shrestha I, Vazquez A, Wendelborn J, Jimenez V, Lisha N, Neilands TB, Scott H, Liu A, Steward W, Johnson MO, Saberi P. Improving the HIV PrEP continuum of care using an intervention for healthcare providers: a stepped-wedge study protocol. BMJ Open. 2020 Jul 14;10(7):e040734. doi: 10.1136/bmjopen-2020-040734. PMID 32665393
- [Result] Saberi P, Ming K, Hojilla JC, Scott HM, Neilands TB. HIV Preexposure Prophylaxis in the Time of COVID-19: How a Robust and Responsive HIV Preexposure Prophylaxis Intervention Can Avert Loss of HIV Prevention Coverage During a Global Pandemic. J Acquir Immune Defic Syndr. 2021 May 1;87(1):e173-e176. doi: 10.1097/QAI.0000000000002652. No abstract available. PMID 33534275
- See also: Related Info — https://prep.ucsf.edu/